CLINICAL TRIAL: NCT02146014
Title: Effects of Transcranial Direct Current Stimulation of the Prefrontal Cortex on Cigarette Smoking
Brief Title: Effects of Transcranial Direct Current Stimulation on Cigarette Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Joaquim Brasil-Neto, Dr., University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAB-69168
Record Dates: First submitted 2014-05-13; First posted 2014-05-23 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Addiction
Keywords: cigarette smoking, smoking
MeSH Terms: conditions — Behavior, Addictive; Cigarette Smoking | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Direct Current Stimulation (Experimental): These subjects will receive real transcranial direct current stimulation.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS (Placebo Comparator): These subjects will receive sham transcranial direct current stimulation (placebo)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Transcranial Direct Current Stimulation (tDCS) is a procedure that uses a small battery-driven unit to deliver weak electrical currents (1-2 mA) through the intact scalp. The procedure is painless and is thought to modulate the excitability of the underlying cerebral tissue for hours or days after sessions.
  In the placebo group the current will be off.
  Arms: Sham tDCS
Device: Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation (tDCS) is a procedure that uses a small battery-driven unit to deliver weak electrical currents (1-2 mA) through the intact scalp. The procedure is painless and is thought to modulate the excitability of the underlying cerebral tissue for hours or days after sessions.
  Arms: Transcranial Direct Current Stimulation

SUMMARY:
Tobacco addiction is treatable with behavioral and pharmacological means, but results are often less than optimal. Transcranial direct current stimulation is a new non-invasive technique that applies weak electrical currents through the skull and has been shown to alter the excitability of certain brain areas. It is currently being tried in disorders where there is abnormal brain excitability, such as epilepsy and depression. A few studies have also been able to diminish drug craving, suggesting that brain excitability might also be altered in drug addiction.

This study aims at non-invasively changing the excitability of certain brain areas-a procedure called neuromodulation- in order to help smokers quit smoking more easily.

ELIGIBILITY:
Inclusion Criteria:

* smokers

Exclusion Criteria:

* use of psychoactive drugs
* age above 70

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analogue Scale of Cigarette Craving | Before and 7 days after treatment

SECONDARY OUTCOMES:
Change in Visual Analogue Scale of Motivation to Quit Smoking | Before and 7 days after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Boechat-Barros, MD, Principal Investigator — University of Brasilia
Locations (1):
- Hospital Universitário de Brasília- HUB, Brasília, Federal District, Brazil

REFERENCES:
- [Derived] Vitor de Souza Brangioni MC, Pereira DA, Thibaut A, Fregni F, Brasil-Neto JP, Boechat-Barros R. Effects of Prefrontal Transcranial Direct Current Stimulation and Motivation to Quit in Tobacco Smokers: A Randomized, Sham Controlled, Double-Blind Trial. Front Pharmacol. 2018 Jan 26;9:14. doi: 10.3389/fphar.2018.00014. eCollection 2018. PMID 29434547